CLINICAL TRIAL: NCT01624389
Title: Establish Taiwan Alzheimer's Disease Neuroimaging Initiative - a Three-year Pilot Study
Acronym: Alzheimer's
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 101-1074A1
Record Dates: First submitted 2012-06-17; First posted 2012-06-20 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-01

CONDITIONS: Alzheimer's Disease
Keywords: [18F]AV-45 PET amyloid binding imaging; Alzheimer's disease
MeSH Terms: conditions — Alzheimer Disease | interventions — florbetapir

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- F18-AV45 (Experimental)
  Interventions: Drug: F18-AV45

INTERVENTIONS:
Drug: F18-AV45 — This study will recruit a total of 200 evaluable subjects (50 cognitively normal volunteers, 100 MCI, and 50 AD, respectively) Each evaluable subject involved in this study must fulfill all the inclusion and exclusion criteria according the subject grouping.
  Safety measurement will be evaluated by medical history, vital signs, physical examinations, laboratory examinations and collecting of adverse events.

SUMMARY:
Alzheimer's disease (AD) may be one of the most pressing problems facing all countries around the world as the population ages.AD is a slowly evolving process that likes begins years to decades before the clinical symptoms area manifest. However, as one would like to identify the disease process at an earlier point in the clinical continuum, the precision of the diagnosis is reduced. Therefore, the challenge is to try to identify the process at the pre-dementia stage and enhance the specificity of the clinical diagnosis through the use of imaging and other biomarkers. Mild cognitive impairment (MCI) represents an attempt to characterize subjects at an early clinical phase of AD and subjects with MCI have been a target for prevention trials. There are two pathological landmarks, in terms of extra-cellular senile plaques and intracellular neurofibrillary tangles. Although present symptomatic treatments provide some benefit to patients with AD, they are not the solution for AD. Up to date, there are still no therapies can alter the underlying nature of the AD process. Therefore, the earlier the intervention takes place, presumably, the greater the protection against further neuronal damage will be appreciated.The Alzheimer's Disease Neuroimaging Initiate (ADNI) is a consortium of universities and medical centers in the United States and Canada established to develop standardized imaging techniques and biomarkers procedures in normal subjects, subjects with MCI and subjects with mild AD. ADNI has been a groundbreaking project, establishing pre-competitive collaboration and real-time data sharing among academia and industry investigators to clarify the relationships among demographic, genetic, clinical, cognitive, neuroimaging and biochemical measures throughout the course of AD neurobiology, in order to facilitate the development of effective therapeutics.This project has exceeded expectations, providing insights into disease mechanisms as well as hugely valuable advances, based primarily on the use of standardized biomarkers, to drug development programs. A number of the leading disease-modifying drug development programs are now employing ADNI methodology toward more efficient trial design, particularly in the critically important early (pre-dementia) AD population

DETAILED DESCRIPTION:
Eligibility:

1. Normal subjects: MMSE scores between 24-30 (inclusive), a CDR of 0, non-depressed, non-MCI, and nondemented, education adjusted scores on Wechsler Memory Scale Logical Memory III story A delayed recall scores (education ≥16 years:≥9; 6-15 years: ≥5).
2. EMCI subjects: MMSE scores between 24-30(inclusive), a memory complaint, have objective memory loss measured by education adjusted scores on Wechsler Memory Scale Logical Memory III story A delayed recall scores (education ≥16 years: 9-11; 6-15 years: 5-9), a CDR sum of box of 0.5 (0.5 only in memory subdomain), absence of significant levels of impairment in other cognitive domains, essentially preserved activities of daily living, and an absence of dementia.
3. LMCI subjects: MMSE scores between 24-30(inclusive), a memory complaint, have objective memory loss measured by education adjusted scores on Wechsler Memory Scale Logical Memory III story A delayed recall scores (education ≥16 years: ≤8; 6-15 years: ≤4), a CDR of 0.5 with a mandatory requirement of the memory box score being 0.5 or greater, essentially preserved activities of daily living, and an absence of dementia.

ELIGIBILITY:
Inclusion Criteria:

Enrolled subjects will be between 55-90 (inclusive) years of age, at least 6 years of formal education, and have a study partner able to provide an independent evaluation of functioning. All subjects must be willing and able to undergo all test procedures including neuroimaging and agree to longitudinal follow up. Specific psychoactive medications will be excluded. General inclusion/exclusion criteria are as follows:

1. Normal subjects: MMSE scores between 24-30 (inclusive), a CDR of 0, non-depressed, non-MCI, and nondemented, education adjusted scores on Wechsler Memory Scale Logical Memory III story A delayed recall scores (education ≥16 years:≥9; 6-15 years: ≥5).
2. EMCI subjects: MMSE scores between 24-30(inclusive), a memory complaint, have objective memory loss measured by education adjusted scores on Wechsler Memory Scale Logical Memory III story A delayed recall scores (education ≥16 years: 9-11; 6-15 years: 5-9), a CDR sum of box of 0.5 (0.5 only in memory subdomain), absence of significant levels of impairment in other cognitive domains, essentially preserved activities of daily living, and an absence of dementia.
3. LMCI subjects: MMSE scores between 24-30(inclusive), a memory complaint, have objective memory loss measured by education adjusted scores on Wechsler Memory Scale Logical Memory III story A delayed recall scores (education ≥16 years: ≤8; 6-15 years: ≤4), a CDR of 0.5 with a mandatory requirement of the memory box score being 0.5 or greater, essentially preserved activities of daily living, and an absence of dementia.
4. Mild AD: MMSE scores between 20-26 (inclusive), CDR of 0.5 or 1.0, and meets NINCDS/ADRDA criteria for probable AD, have objective memory loss measured by education adjusted scores on Wechsler Memory Scale Logical Memory III story A delayed recall scores (education ≥16 years: ≤8; 6-15 years: ≤4)

Exclusion criteria:

Subjects taking antidepressant medications with anticholinergic properties will be excluded, and the regular use of narcotic agents have to be limited to < 2 doses per week within 4 weeks of screening. Neuroleptic medications and other drugs with anticholinergic properties, anti-parkinsonian medications are not allowed within 4 weeks of screening. Diuretic drugs should not be started or need to be discontinued 4 weeks prior to screening. Cholinesterase inhibitors and memantine are permitted if the doses are stable for 4 weeks prior to screening for subjects with MCI and AD. Estrogen and estrogen-like compounds and vitamin E are allowed if the dose have been stable for 4 weeks prior to screening. Participants are required to report any medication changes to the site investigators once they are enrolled in the study.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-01; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Rate of conversion from NC, EMCI, LMCI to AD. | three years

CONTACTS AND LOCATIONS:
Overall Officials: Tzu-Chen YEN, MD,PhD, Study Director — Nuclear Medicine
Locations (1):
- Tzu-Chen-Yen, Taoyuan District, Taiwan